CLINICAL TRIAL: NCT07056478
Title: RANKL Inhibition to Combat Sarcopenia in Hip Fracture Patients: A Pragmatic, Randomized Double-blind, Active-Controlled Trial
Brief Title: RANKL Inhibition to Combat Sarcopenia in Hip Fracture Patients
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Prince of Wales Hospital, Shatin, Hong Kong (Other)
Responsible Party: Principal Investigator, Ronald Man Yeung WONG, Clinical Associate Professor, Prince of Wales Hospital, Shatin, Hong Kong
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2023.401
Record Dates: First submitted 2025-06-19; First posted 2025-07-09 (Actual); Last update posted 2025-07-09 (Actual); Status verified 2025-06

CONDITIONS: Sarcopenia in Elderly
MeSH Terms: interventions — Denosumab; Zoledronic Acid

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Denosumab group (Active Comparator): 60mg subcutaneous Denosumab (1mL solution) every 6 months and intravenous placebo (100mL normal saline) once yearly
  Interventions: Drug: Denosumab (Prolia)
- Zolendronic acid group (Placebo Comparator): 5mg intravenous Zoledronic Acid (100mL solution) once yearly and subcutaneous placebo (1mL normal saline) every 6 months
  Interventions: Drug: Zoledronic acide (Aclasta)

INTERVENTIONS:
Drug: Denosumab (Prolia) — 60mg subcutaneous Denosumab (1mL solution) every 6 months and intravenous placebo (100mL normal saline) once yearly
  Arms: Denosumab group
Drug: Zoledronic acide (Aclasta) — 5mg intravenous Zoledronic Acid (100mL solution) once yearly and subcutaneous placebo (1mL normal saline) every 6 months
  Arms: Zolendronic acid group

SUMMARY:
The objective of this study is to conduct a pragmatic, randomized, double-blind, active-controlled trial to assess the efficacy of receptor activator of nuclear factor-kB ligand (RANKL) inhibition in the treatment of sarcopenia in hip fractures.

DETAILED DESCRIPTION:
Objectives

1. To investigate the effect of RANKL inhibition in treating sarcopenia in hip fracture patients in terms of physical performance and quality of life.
2. To investigate the effect of RANKL inhibition in treating sarcopenia in hip fracture patients in terms of appendicular skeletal muscle mass and muscle strength.
3. To investigate the efficacy of RANKL inhibition in treating sarcopenia in hip fracture patients in terms of falls, hospital re-admissions, re-fractures, and mortality.

ELIGIBILITY:
Inclusion Criteria:

* Elderly aged 65 years or older
* Diagnosed with sarcopenia following AWGS guidelines - low appendicular skeletal muscle mass measured by dual-energy x-ray absorptiometry (Cutoff: Male <7.0kg/m2, and female <5.4kg/m2) AND low handgrip strength (Cutoff: Male < 28kg, Female <18 kg) OR low physical performance (6-metre walk, cutoff: <1.0m/s or 5-time chair stand test >=12s)
* Diagnosed with a hip fracture from low-energy mechanism (e.g., falling from standing height) requiring an operation
* Willing and able to comply with study protocol including follow-up evaluations.

Exclusion Criteria:

* open fracture
* multiple fractures
* pathological fractures e.g., tumour, infection, etc.
* history of medication or disease affecting bone metabolism e.g., hypo/hyperthyroidism
* malignancy
* chairbound or bedbound (unable to perform assessments)
* serious cognitive problems e.g., severe dementia (unable to agree for consent) - renal impairment with glomerular filtration rate <30 mL/min
* prior anti-osteoporotic medication e.g. bisphosphonates, denosumab, etc.
* active infection,
* severe malnutrition i.e. Mini Nutritional Assessment < 17 points
* serious neurological or neuromuscular conditions e.g. Parkinson's disease
* uncontrolled chronic conditions e.g. poorly controlled diabetes mellitis
* not anaesthetically fit for operation or conservative management

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 130 (Estimated)
Dates: Start 2026-01-01 (Estimated); Primary Completion 2028-01-01 (Estimated); Study Completion 2030-01-01 (Estimated)

PRIMARY OUTCOMES:
Sarcopenia and Quality of Life (SarQoL®) | From enrolment to 24 months after the start of treatment
  Health-related questionnaire for sarcopenia which is composed of 55 items translated into 22 questions and organized into seven domains of quality of life including physical and mental health, locomotion, body composition, functionality, activities of daily living, leisure activities, and fears. The SarQoL involves an overall score, which is the sum of seven individual domain scores, with higher scores indicating better quality of life. During the scoring process, the overall and domain scores are rescaled such that their maximum possible values become 100.
Quadriceps muscle strength | From enrolment to 24 months after the start of treatment
  Measured on affected limb with isometric dynamometer (Baseline, Genova, Italy). Subject will sit on a chair with both feet above ground, while raising the affected leg 45° forwards. The dynamometer is placed above the ankle and subject will push the leg forward with maximum force. Measurements are repeated three times and maximum value used for evaluation
Handgrip strength | From enrolment to 24 months after the start of treatment
  Assessed by handgrip strength with spring-type hand dynamometer (JAMAR Hand Dynamometer 5030JO; Sammons Preston, Bolingbrook, IL). The maximum reading of 2 trials using the dominant hand in a maximum-effort isometric contraction is taken. Male < 28kg, and female <18kg are cut-off for low handgrip strength
Appendicular skeletal muscle mass (ASM) | From enrolment to 24 months after the start of treatment
  Determined with Dual-energy X-ray absorptiometry (Horizon®, Hologic, USA). Total appendicular skeletal mass (ASM) is evaluated by segmented measurement of muscle mass at four limbs by operator-defined cutlines at specific anatomical landmarks. ASM is adjusted to square of height to calculate appendicular skeletal mass index (ASMI) (kg/m2). Cutoff of low ASMI is defined as Male <7.0kg/m2, and female <5.4kg/m2.
5-time chair stand test | From enrolment to 24 months after the start of treatment
  The time to rise from a chair 5 times is recorded. Low physical performance is ≥ 12 seconds.
6-metre walk | From enrolment to 24 months after the start of treatment
  The time taken to walk 6 metres without deceleration is taken. The average result of 2 trials is taken and recorded. Low physical performance is <1.0m/s
Short Physical Performance Battery | From enrolment to 24 months after the start of treatment
  Performed by balance test (side-by-side stand, semi-tandem stand, and tandem stand), gait speed test (time for 4-meter walk), and chair stand test (5 repeats). Low physical performance is ≤ 9.
Balancing ability | From enrolment to 24 months after the start of treatment
  The Basic Balance Master System (NeuroCom International Inc, USA) is used to measure static and dynamic ability of subjects to maintain center of balance. Subjects will stand barefoot on force plate and control location of their center-of-gravity by weight-shifting to eight different targets. Measured parameters of limits of stability test includes reaction time(s).
Balancing ability | From enrolment to 24 months after the start of treatment
  The Basic Balance Master System (NeuroCom International Inc, USA) is used to measure static and dynamic ability of subjects to maintain center of balance. Subjects will stand barefoot on force plate and control location of their center-of-gravity by weight-shifting to eight different targets. Measured parameters of limits of stability test includes directional control (%).
Balancing ability | From enrolment to 24 months after the start of treatment
  The Basic Balance Master System (NeuroCom International Inc, USA) is used to measure static and dynamic ability of subjects to maintain center of balance. Subjects will stand barefoot on force plate and control location of their center-of-gravity by weight-shifting to eight different targets. Measured parameters of limits of stability test includes movement velocity (degrees/s).
Balancing ability | From enrolment to 24 months after the start of treatment
  The Basic Balance Master System (NeuroCom International Inc, USA) is used to measure static and dynamic ability of subjects to maintain center of balance. Subjects will stand barefoot on force plate and control location of their center-of-gravity by weight-shifting to eight different targets. Measured parameters of limits of stability test includes endpoint excursion (%).
Balancing ability | From enrolment to 24 months after the start of treatment
  The Basic Balance Master System (NeuroCom International Inc, USA) is used to measure static and dynamic ability of subjects to maintain center of balance. Subjects will stand barefoot on force plate and control location of their center-of-gravity by weight-shifting to eight different targets. Measured parameters of limits of stability test includes maximum excursion (%).

SECONDARY OUTCOMES:
Falls | From enrolment to 24 months after the start of treatment
  Patients self-report via fall calendar, which will be returned at each follow-up. Calendar reporting has been well proven to be reliable for fall studies
Hospital re-admissions | From enrolment to 24 months after start of treatment
  Documented from Clinical Management System (CMS) from Hospital Authority (public computerized system for all patients)
Secondary fracture | From enrolment to 24 months after start of treatment
  Confirmed via X-ray/radiology report and Clinical Management System (CMS). Lateral X-ray of spine also taken during follow-up to detect the often clinically silent vertebral fracture. Vertebra is assessed by Genant classification as per our previously established protocol
Mortality | From enrolment to 24 months after start of treatment
  Documented from the Clinical Management System (CMS) from Hospital Authority (public computerized system for all patients)
Bone mineral density (BMD) | From enrolment to 24 months after the start of treatment
  Measured by Dual-energy X-ray absorptiometry (Horizon®, Hologic, US) at lumbar spine and contralateral hip

CONTACTS AND LOCATIONS:
Locations (1):
- The Chinese University of Hong Kong, Hong Kong, China

IPD SHARING:
Plan to Share IPD: No